CLINICAL TRIAL: NCT04630132
Title: Renal Ageing-sarcopenia Network: a Combined Genetic, Immunological and Psychological Approach to Dissect Frailty
Brief Title: Renal Ageing-sarcopenia Network
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Cariplo Foundation (Unknown)
Responsible Party: Principal Investigator, Paolo Manunta, Professor, IRCCS San Raffaele
Other Study IDs: FRASNET
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Aging; Frailty; Hypertension; CKD
Keywords: aging; Klotho; Hypertension; physical activity; frailty; sarcopenia; body composition; CKD; cognitive impairment; depression; inflammation; citokine; adducin; ouabain
MeSH Terms: conditions — Frailty; Hypertension; Motor Activity; Sarcopenia; Cognitive Dysfunction; Depression; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frailty Group: The 'phenotype' of frailty (cases) is defined as follows: presence of three or more of the following features:
  1. Decreased grip strength
  2. Self-reported exhaustion
  3. Unintentional weight loss of more than 4.5 kg over the past year
  4. Slow walking speed
  5. Low physical activity
- Non-Frailty Group: The 'phenotype' of non-frailty (control) is defined as follows: presence of less than three of the following features:
  1. Decreased grip strength
  2. Self-reported exhaustion
  3. Unintentional weight loss of more than 4.5 kg over the past year
  4. Slow walking speed
  5. Low physical activity

SUMMARY:
Frailty is a syndrome in which the accumulation of small, individually insignificant deficits leads to heightened vulnerability to adverse events and predisposes to potential catastrophic decompensation.

Objective of this study is to clarify the underlying genetic and immunological mechanisms responsible of frailty condition focused on: i. nephrosclerosis ageing kidney phenotype related to salt effects on immunosystem, ii. immunological aspect of sarcopenia, iii. psychological disorder related to immunosystem activation, iv. detection of new biomarkers of frailty.

DETAILED DESCRIPTION:
The cross-sectional, observational cohort study include 1500 subjects (age >65 years) subdivided in 750 cases and 750 controls according to frailty.

Subjects who met the following criteria are included: 1) older than 65; 2) able to walk 500 m without assistance; 3) a Mini-Mental State Examination (MMSE) score <18; and 4) no severe health problems (eg, uncontrolled hypertension, recent upper or lower extremity fractures, myocardial infarction within the past 1 year).

According to definition for the 'phenotype' of frailty (cases) is as follows: presence of three or more of the following features:

1. Decreased grip strength
2. Self-reported exhaustion
3. Unintentional weight loss of more than 4.5 kg over the past year
4. Slow walking speed
5. Low physical activity

The investigators select as control subjects with presence of less than 1 criteria . All the control subjects are evaluated by the same protocol than the cases. Subjects will be collected in collaboration with senior housing (RSA) of Milano city, country clubs, social club for elderly, and elderly university. The study will be approved by the Ethics Committee of ASL of Milano city and at individual centers by local ethical committees. All the study participants signed informed consent. At the baseline evaluation, a large amount of data is collected. First, the participants completed a battery of self-reported questionnaires concerning the demographic characteristics, psychosocial adjustment, quality of life, and health condition, in the presence of a trained psychologist in order to clarify any doubts. Second, an expert in physical education and adapted physical activity for older adults administered physical tests. Finally, people with expertise in the eld of ergonomics take anthropometric measurements. Data collection is always carried out in the same order and individually for each participant.

In all the subjects following clinical and laboratoristic data are collected:

1. Clinical evaluation:

1. Collection of anamnestic data.
2. Blood pressure measurement. Blood pressure is measured by a trained nurse using an authomatic device (OMRON) and an appropriately sized cuff. Readings are obtained after 5 min of seated rest. The mean of 3 blood pressure measurements obtained at 1-min intervals during the medical evaluation is used to define SBP and DBP.
3. Evaluation of kidney function :

   a. CKD is defined as a glomerular filtration rate (GFR) lower than 60 mL/min/1.73 m2 or markers of kidney damage, such as albuminuria,for greater than 3 months. A creatinine-based formula is used to estimate GFR, applying Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equations.

   b. Urine analysis and albumin /creatinine and sodium /creatinine ratio urinary excretion.

2. Physical frailty measure. To identify physically frail older adults, an adapted version of the frailty phenotype of Fried et al is used. Subjects with three or more criteria are classified as frail, those with one or two as prefrail, and those meeting none as robust.

1. Body composition: Height and weight are detected. Bioimpedance analysis (BIA) is a system of evaluation of body composition, able to calculate adjunctive information: total body water (TBW), extra and intracellular water (ECW and ICW), body cell mass (BCM), muscle mass (MM), fat mass (FM), fat free mass (FFM), basal metabolic rate.
2. SPPB: The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance).
3. PASE: Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of persons age 65 years and older. The PASE score combines information on leisure, household and occupational activity. The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.

Sarcopenia will be defined as fat-free mass index (FFMI) below the 25th percentile combined with one of the following functional parameter: either an SPPB score ≤8 or a comfortable gait speed <1.0 m/s.

3. Psychological test will be used to assess self conditions

1. Mini Mental State Examination (MMSE): The Mini-Mental Stat Examination (MMSE) is a 10-minute measure of cognitive impairment in undeveloped, uneducated, diseased, or very old populations.
2. Geriatric Depression Scale-short form (GDS-15): The Geriatric Depression Scale (GDS) is a 15- item self-report validated measure for rating depression in elderly adults. Additionally, the GDS is sensitive to depression among elderly adults suffering from mild to moderate dementia and elderly adults with physical illnesses by excluding questions pertaining to somatic complaints and cognitive dimension of depression. In this scale, a score of 6 or higher may be indicative of depression and must be evaluated jointly with patient's clinical data.
3. SF-36 Medical Outcomes Study (MOS) 36-item Short Form Health Survey: This instrument should capture both mental and physical aspects of health. The 36 6-likert item assess health across eight domains, namely bodily pain, general health perceptions, mental health, physical functioning, role limitations due to emotional health problems, role limitations due to physical health problems, social functioning, and vitality. All items use categorical response options (range: 2-6 options). Two component summary scores for physical and mental health (MPS and MCS, respectively) can also be calculated.

4. Laboratory Methods

1. Genotyping. OpenArray technology (ThermoFisher) for genetic characterization of Single Nucleotide Polymorphisms (SNPs), based on TaqMan chemistry. DNA will be used for genotyping of genetic variants in loci for Klotho (KL) gene, Adducins (ADD1, ADD2 and ADD3) and EO synthesis (LSS, HSD3B1), metabolism (CYP11A1, ABCB1), and activity (SLC8A1, SIK1) genes, and for immunological pathway (TLR4, HMGB1, IL6, IL1).
2. Biochemical measurements.

   1. Endogenous Ouabain measurement
   2. Plasma Klotho measurement.
3. Immunological determinations. Simultaneous assessment of serum concentrations of epidermal growth factor (EGF), fibroblast growth factor 2 (FGF2), FMS-like tyrosine kinase 3 ligand (Flt-3L), granulocyte colony-stimulating factor (G-CSF), granulocyte-monocyte colonystimulating factor (GM-CSF), interferon-α2 (IFN-α2), INF-γ, IL-10, IL-15, IL-17, IL-1β, IL-2, IL-6, IL-8, INF-γ inducible protein 10 (IP-10), monocyte chemoattractant protein-1 (MCP-1), macrophage inflammatory protein-1β (MIP-1 β), platelet-derived growth factor-AA (PDGF-AA), soluble CD40 ligand (sCD40L), transforming growth factor alpha (TGF-α), TNF-α and vascular endothelial growth factor (VEGF).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Male and female patients
* Patients able to walk > 500 m without assistance
* MMSE < 18
* No severe health problems (Uncontrolled hypertension, recent upper or lower extremity fractures, myocardial infarction within the past 1 year).

Exclusion Criteria:

* Severe cardiological or pulmonary disease (NYHA IV, Gold IV)
* Intracranial interventions
* Dying patients (palliative situation)
* Not enough language skills
* Non-consenting patients
* Participation in another prospective intervention study for study inclusion or throughout the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community sample of the elderly population
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-03-25 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between Frailty and Klotho polymorphism, assessed by Fried Classification: non-frail (score 0), pre-frail (score 1-2) and frail (score 3-5) | 3 years
  Verifying the role of the polymorphism of the Klotho gene in the development of the "fragility" phenotype in elderly subjects.

SECONDARY OUTCOMES:
Correlation between Frailty and Klotho (KL), Adducine (ADD1, ADD2 and ADD3), Lanosterol and other polymorphisms, assessed by Fried Classification: non-frail (score 0), pre-frail (score 1-2) and frail (score 3-5) | 3 years
  Finding genetic profiles predisposing to the development of frailty through genotyping for Klotho (KL), Adducine (ADD1, ADD2 and ADD3), Lanosterol and further polymorphisms in genes related to renal function and the immune system.
Correlation between Frailty and plasmatic values of endogenous ouabain, Klotho and plasma cytokines, assessed by Fried Classification: non-frail (score 0), pre-frail (score 1-2) and frail (score 3-5) | 3 years
  Studying the role of biomarkers in the development of frailty: endogenous ouabain, Klotho and plasma cytokines.
Creation of a multidisciplinary frailty score, based on the outcomes of the study | 3 years
  Building a multidisciplinary frailty score based on biochemical, genetic and psychological results of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Manunta, PhDMD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Clinical data and sample alredy collectd are available,

REFERENCES:
- [Background] Barabasi AL, Gulbahce N, Loscalzo J. Network medicine: a network-based approach to human disease. Nat Rev Genet. 2011 Jan;12(1):56-68. doi: 10.1038/nrg2918. PMID 21164525
- [Background] Barabasi AL. Network medicine--from obesity to the "diseasome". N Engl J Med. 2007 Jul 26;357(4):404-7. doi: 10.1056/NEJMe078114. Epub 2007 Jul 25. No abstract available. PMID 17652657
- [Background] Goh KI, Cusick ME, Valle D, Childs B, Vidal M, Barabasi AL. The human disease network. Proc Natl Acad Sci U S A. 2007 May 22;104(21):8685-90. doi: 10.1073/pnas.0701361104. Epub 2007 May 14. PMID 17502601
- [Background] Kyle UG, Genton L, Hans D, Karsegard VL, Michel JP, Slosman DO, Pichard C. Total body mass, fat mass, fat-free mass, and skeletal muscle in older people: cross-sectional differences in 60-year-old persons. J Am Geriatr Soc. 2001 Dec;49(12):1633-40. doi: 10.1046/j.1532-5415.2001.t01-1-49272.x. PMID 11843996
- [Background] Melton LJ 3rd, Riggs BL, Achenbach SJ, Amin S, Camp JJ, Rouleau PA, Robb RA, Oberg AL, Khosla S. Does reduced skeletal loading account for age-related bone loss? J Bone Miner Res. 2006 Dec;21(12):1847-55. doi: 10.1359/jbmr.060908. PMID 17002566
- [Background] Newman AB, Haggerty CL, Goodpaster B, Harris T, Kritchevsky S, Nevitt M, Miles TP, Visser M; Health Aging And Body Composition Research Group. Strength and muscle quality in a well-functioning cohort of older adults: the Health, Aging and Body Composition Study. J Am Geriatr Soc. 2003 Mar;51(3):323-30. doi: 10.1046/j.1532-5415.2003.51105.x. PMID 12588575
- [Background] Morley JE, Anker SD, von Haehling S. Prevalence, incidence, and clinical impact of sarcopenia: facts, numbers, and epidemiology-update 2014. J Cachexia Sarcopenia Muscle. 2014 Dec;5(4):253-9. doi: 10.1007/s13539-014-0161-y. Epub 2014 Oct 22. PMID 25425503
- [Background] Abellan van Kan G. Epidemiology and consequences of sarcopenia. J Nutr Health Aging. 2009 Oct;13(8):708-12. doi: 10.1007/s12603-009-0201-z. PMID 19657554
- [Background] Janssen I. The epidemiology of sarcopenia. Clin Geriatr Med. 2011 Aug;27(3):355-63. doi: 10.1016/j.cger.2011.03.004. Epub 2011 May 14. PMID 21824552
- [Background] Liu CK, Leng X, Hsu FC, Kritchevsky SB, Ding J, Earnest CP, Ferrucci L, Goodpaster BH, Guralnik JM, Lenchik L, Pahor M, Fielding RA. The impact of sarcopenia on a physical activity intervention: the Lifestyle Interventions and Independence for Elders Pilot Study (LIFE-P). J Nutr Health Aging. 2014 Jan;18(1):59-64. doi: 10.1007/s12603-013-0369-0. PMID 24402391
- [Background] Muscaritoli M, Lucia S, Molfino A. Sarcopenia in critically ill patients: the new pandemia. Minerva Anestesiol. 2013 Jul;79(7):771-7. Epub 2013 Jan 31. PMID 23370125
- [Background] Kalinkovich A, Livshits G. Sarcopenia--The search for emerging biomarkers. Ageing Res Rev. 2015 Jul;22:58-71. doi: 10.1016/j.arr.2015.05.001. Epub 2015 May 8. PMID 25962896
- [Background] Glassock RJ, Rule AD: The kidney in aging. In Davison AM, Cameron S, Grunfeld J-P, Ponticelli C (eds): Oxford Textbook of Clinical Nephrology, ed. 3, Oxford, Oxford University press, (2015
- [Background] Glassock RJ, Rule AD. The implications of anatomical and functional changes of the aging kidney: with an emphasis on the glomeruli. Kidney Int. 2012 Aug;82(3):270-7. doi: 10.1038/ki.2012.65. Epub 2012 Mar 21. PMID 22437416
- [Background] Wang X, Vrtiska TJ, Avula RT, Walters LR, Chakkera HA, Kremers WK, Lerman LO, Rule AD. Age, kidney function, and risk factors associate differently with cortical and medullary volumes of the kidney. Kidney Int. 2014 Mar;85(3):677-85. doi: 10.1038/ki.2013.359. Epub 2013 Sep 25. PMID 24067437
- [Background] Roeder SS, Stefanska A, Eng DG, Kaverina N, Sunseri MW, McNicholas BA, Rabinovitch P, Engel FB, Daniel C, Amann K, Lichtnekert J, Pippin JW, Shankland SJ. Changes in glomerular parietal epithelial cells in mouse kidneys with advanced age. Am J Physiol Renal Physiol. 2015 Jul 15;309(2):F164-78. doi: 10.1152/ajprenal.00144.2015. Epub 2015 May 27. PMID 26017974
- [Background] Shankland SJ, Anders HJ, Romagnani P. Glomerular parietal epithelial cells in kidney physiology, pathology, and repair. Curr Opin Nephrol Hypertens. 2013 May;22(3):302-9. doi: 10.1097/MNH.0b013e32835fefd4. PMID 23518463
- [Background] Mekli K, Marshall A, Nazroo J, Vanhoutte B, Pendleton N. Genetic variant of Interleukin-18 gene is associated with the Frailty Index in the English Longitudinal Study of Ageing. Age Ageing. 2015 Nov;44(6):938-42. doi: 10.1093/ageing/afv122. Epub 2015 Sep 22. PMID 26396182
- [Background] Tripodi G, Citterio L, Kouznetsova T, Lanzani C, Florio M, Modica R, Messaggio E, Hamlyn JM, Zagato L, Bianchi G, Staessen JA, Manunta P. Steroid biosynthesis and renal excretion in human essential hypertension: association with blood pressure and endogenous ouabain. Am J Hypertens. 2009 Apr;22(4):357-63. doi: 10.1038/ajh.2009.3. Epub 2009 Feb 5. PMID 19197249
- [Background] Manunta P, Messaggio E, Casamassima N, Gatti G, Carpini SD, Zagato L, Hamlyn JM. Endogenous ouabain in renal Na(+) handling and related diseases. Biochim Biophys Acta. 2010 Dec;1802(12):1214-8. doi: 10.1016/j.bbadis.2010.03.001. Epub 2010 Mar 11. PMID 20226856
- [Background] Citterio L, Lanzani C, Manunta P, Bianchi G. Genetics of primary hypertension: the clinical impact of adducin polymorphisms. Biochim Biophys Acta. 2010 Dec;1802(12):1285-98. doi: 10.1016/j.bbadis.2010.03.014. Epub 2010 Apr 8. PMID 20382219
- [Background] Chen X, Mao G, Leng SX. Frailty syndrome: an overview. Clin Interv Aging. 2014 Mar 19;9:433-41. doi: 10.2147/CIA.S45300. eCollection 2014. PMID 24672230
- [Background] Wade B, Abais-Battad JM, Mattson DL. Role of immune cells in salt-sensitive hypertension and renal injury. Curr Opin Nephrol Hypertens. 2016 Jan;25(1):22-7. doi: 10.1097/MNH.0000000000000183. PMID 26575395
- [Background] Guzik TJ, Hoch NE, Brown KA, McCann LA, Rahman A, Dikalov S, Goronzy J, Weyand C, Harrison DG. Role of the T cell in the genesis of angiotensin II induced hypertension and vascular dysfunction. J Exp Med. 2007 Oct 1;204(10):2449-60. doi: 10.1084/jem.20070657. Epub 2007 Sep 17. PMID 17875676
- [Background] Youn JC, Yu HT, Lim BJ, Koh MJ, Lee J, Chang DY, Choi YS, Lee SH, Kang SM, Jang Y, Yoo OJ, Shin EC, Park S. Immunosenescent CD8+ T cells and C-X-C chemokine receptor type 3 chemokines are increased in human hypertension. Hypertension. 2013 Jul;62(1):126-33. doi: 10.1161/HYPERTENSIONAHA.113.00689. Epub 2013 May 28. PMID 23716586
- [Background] Kuro-o M. Klotho and aging. Biochim Biophys Acta. 2009 Oct;1790(10):1049-58. doi: 10.1016/j.bbagen.2009.02.005. Epub 2009 Feb 20. PMID 19230844
- [Background] Wang Y, Sun Z. Current understanding of klotho. Ageing Res Rev. 2009 Jan;8(1):43-51. doi: 10.1016/j.arr.2008.10.002. Epub 2008 Oct 31. PMID 19022406
- [Background] Di Bona D, Accardi G, Virruso C, Candore G, Caruso C. Association of Klotho polymorphisms with healthy aging: a systematic review and meta-analysis. Rejuvenation Res. 2014 Apr;17(2):212-6. doi: 10.1089/rej.2013.1523. Epub 2014 Apr 11. PMID 24164579
- [Background] Mengel-From J, Soerensen M, Nygaard M, McGue M, Christensen K, Christiansen L. Genetic Variants in KLOTHO Associate With Cognitive Function in the Oldest Old Group. J Gerontol A Biol Sci Med Sci. 2016 Sep;71(9):1151-9. doi: 10.1093/gerona/glv163. Epub 2015 Sep 24. PMID 26405063
- [Background] Shardell M, Semba RD, Rosano C, Kalyani RR, Bandinelli S, Chia CW, Ferrucci L. Plasma Klotho and Cognitive Decline in Older Adults: Findings From the InCHIANTI Study. J Gerontol A Biol Sci Med Sci. 2016 May;71(5):677-82. doi: 10.1093/gerona/glv140. Epub 2015 Aug 21. PMID 26297657
- [Background] Hsu YH, Liang CK, Chou MY, Liao MC, Lin YT, Chen LK, Lo YK. Association of cognitive impairment, depressive symptoms and sarcopenia among healthy older men in the veterans retirement community in southern Taiwan: a cross-sectional study. Geriatr Gerontol Int. 2014 Feb;14 Suppl 1:102-8. doi: 10.1111/ggi.12221. PMID 24450567
- [Background] Bremmer MA, Beekman AT, Deeg DJ, Penninx BW, Dik MG, Hack CE, Hoogendijk WJ. Inflammatory markers in late-life depression: results from a population-based study. J Affect Disord. 2008 Mar;106(3):249-55. doi: 10.1016/j.jad.2007.07.002. Epub 2007 Aug 22. PMID 17716746
- [Background] Penninx BW, Kritchevsky SB, Yaffe K, Newman AB, Simonsick EM, Rubin S, Ferrucci L, Harris T, Pahor M. Inflammatory markers and depressed mood in older persons: results from the Health, Aging and Body Composition study. Biol Psychiatry. 2003 Sep 1;54(5):566-72. doi: 10.1016/s0006-3223(02)01811-5. PMID 12946885
- [Background] Tiemeier H, Hofman A, van Tuijl HR, Kiliaan AJ, Meijer J, Breteler MM. Inflammatory proteins and depression in the elderly. Epidemiology. 2003 Jan;14(1):103-7. doi: 10.1097/00001648-200301000-00025. PMID 12500057
- [Background] Mulsant BH, Ganguli M. Epidemiology and diagnosis of depression in late life. J Clin Psychiatry. 1999;60 Suppl 20:9-15. PMID 10513852
- [Background] Liu M, Li Y, Citterio L, Huang QF, Zeng WF, Sheng CS, Wei FF, Dong Q, Li GL, Kang YY, Zhang L, Xu TY, Li JJ, Song J, Manunta P, Wang JG. A functional common polymorphism of the ABCB1 gene is associated with chronic kidney disease and hypertension in Chinese. Am J Hypertens. 2013 Dec;26(12):1428-36. doi: 10.1093/ajh/hpt126. Epub 2013 Aug 7. PMID 23926124
- [Background] Licastro F, Pedrini S, Caputo L, Annoni G, Davis LJ, Ferri C, Casadei V, Grimaldi LM. Increased plasma levels of interleukin-1, interleukin-6 and alpha-1-antichymotrypsin in patients with Alzheimer's disease: peripheral inflammation or signals from the brain? J Neuroimmunol. 2000 Feb 1;103(1):97-102. doi: 10.1016/s0165-5728(99)00226-x. PMID 10674995
- [Background] Siu PM, Pistilli EE, Alway SE. Age-dependent increase in oxidative stress in gastrocnemius muscle with unloading. J Appl Physiol (1985). 2008 Dec;105(6):1695-705. doi: 10.1152/japplphysiol.90800.2008. Epub 2008 Sep 18. PMID 18801960
- [Background] Meng SJ, Yu LJ. Oxidative stress, molecular inflammation and sarcopenia. Int J Mol Sci. 2010 Apr 12;11(4):1509-26. doi: 10.3390/ijms11041509. PMID 20480032
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Zuidema S, Koopmans R, Verhey F. Prevalence and predictors of neuropsychiatric symptoms in cognitively impaired nursing home patients. J Geriatr Psychiatry Neurol. 2007 Mar;20(1):41-9. doi: 10.1177/0891988706292762. PMID 17341770
- [Background] Wada T, Ishine M, Sakagami T, Kita T, Okumiya K, Mizuno K, Rambo TA, Matsubayashi K. Depression, activities of daily living, and quality of life of community-dwelling elderly in three Asian countries: Indonesia, Vietnam, and Japan. Arch Gerontol Geriatr. 2005 Nov-Dec;41(3):271-80. doi: 10.1016/j.archger.2005.03.003. Epub 2005 Jun 24. PMID 15979739
- [Background] Strawbridge WJ, Shema SJ, Balfour JL, Higby HR, Kaplan GA. Antecedents of frailty over three decades in an older cohort. J Gerontol B Psychol Sci Soc Sci. 1998 Jan;53(1):S9-16. doi: 10.1093/geronb/53b.1.s9. PMID 9469175
- [Background] Zhou X, Crook MF, Sharif-Rodriguez W, Zhu Y, Ruben Z, Pan Y, Urosevic-Price O, Wang L, Flattery AM, Forrest G, Szeto D, Zhao H, Roy S, Forrest MJ. Chronic antagonism of the mineralocorticoid receptor ameliorates hypertension and end organ damage in a rodent model of salt-sensitive hypertension. Clin Exp Hypertens. 2011;33(8):538-47. doi: 10.3109/10641963.2011.566956. Epub 2011 Sep 27. PMID 21950654
- [Background] Esposito A, Campana L, Palmisano A, De Cobelli F, Canu T, Santarella F, Colantoni C, Monno A, Vezzoli M, Pezzetti G, Manfredi AA, Rovere-Querini P, Del Maschio A. Magnetic resonance imaging at 7T reveals common events in age-related sarcopenia and in the homeostatic response to muscle sterile injury. PLoS One. 2013;8(3):e59308. doi: 10.1371/journal.pone.0059308. Epub 2013 Mar 12. PMID 23555016
- [Background] Georgakis MK, Papadopoulos FC, Protogerou AD, Pagonari I, Sarigianni F, Biniaris-Georgallis SI, Kalogirou EIota, Thomopoulos TP, Kapaki E, Papageorgiou C, Papageorgiou SG, Tousoulis D, Petridou ET. Comorbidity of Cognitive Impairment and Late-Life Depression Increase Mortality: Results From a Cohort of Community-Dwelling Elderly Individuals in Rural Greece. J Geriatr Psychiatry Neurol. 2016 Jul;29(4):195-204. doi: 10.1177/0891988716632913. Epub 2016 Feb 25. PMID 26917554
- [Background] Saracli O, Akca AS, Atasoy N, Onder O, Senormanci O, Kaygisiz I, Atik L. The Relationship between Quality of Life and Cognitive Functions, Anxiety and Depression among Hospitalized Elderly Patients. Clin Psychopharmacol Neurosci. 2015 Aug 31;13(2):194-200. doi: 10.9758/cpn.2015.13.2.194. PMID 26243848
- [Background] Brunelli S, Sciorati C, D'Antona G, Innocenzi A, Covarello D, Galvez BG, Perrotta C, Monopoli A, Sanvito F, Bottinelli R, Ongini E, Cossu G, Clementi E. Nitric oxide release combined with nonsteroidal antiinflammatory activity prevents muscular dystrophy pathology and enhances stem cell therapy. Proc Natl Acad Sci U S A. 2007 Jan 2;104(1):264-9. doi: 10.1073/pnas.0608277104. Epub 2006 Dec 20. PMID 17182743
- [Background] Miglietta D, De Palma C, Sciorati C, Vergani B, Pisa V, Villa A, Ongini E, Clementi E. Naproxcinod shows significant advantages over naproxen in the mdx model of Duchenne Muscular Dystrophy. Orphanet J Rare Dis. 2015 Aug 22;10:101. doi: 10.1186/s13023-015-0311-0. PMID 26296873
- [Background] Touvier T, De Palma C, Rigamonti E, Scagliola A, Incerti E, Mazelin L, Thomas JL, D'Antonio M, Politi L, Schaeffer L, Clementi E, Brunelli S. Muscle-specific Drp1 overexpression impairs skeletal muscle growth via translational attenuation. Cell Death Dis. 2015 Feb 26;6(2):e1663. doi: 10.1038/cddis.2014.595. PMID 25719247
- [Background] Willmann R, De Luca A, Benatar M, Grounds M, Dubach J, Raymackers JM, Nagaraju K; TREAT-NMD Neuromuscular Network. Enhancing translation: guidelines for standard pre-clinical experiments in mdx mice. Neuromuscul Disord. 2012 Jan;22(1):43-9. doi: 10.1016/j.nmd.2011.04.012. Epub 2011 Jul 6. PMID 21737275
- [Background] De Palma C, Morisi F, Cheli S, Pambianco S, Cappello V, Vezzoli M, Rovere-Querini P, Moggio M, Ripolone M, Francolini M, Sandri M, Clementi E. Autophagy as a new therapeutic target in Duchenne muscular dystrophy. Cell Death Dis. 2012 Nov 15;3(11):e418. doi: 10.1038/cddis.2012.159. PMID 23152054
- [Background] De Palma C, Morisi F, Pambianco S, Assi E, Touvier T, Russo S, Perrotta C, Romanello V, Carnio S, Cappello V, Pellegrino P, Moscheni C, Bassi MT, Sandri M, Cervia D, Clementi E. Deficient nitric oxide signalling impairs skeletal muscle growth and performance: involvement of mitochondrial dysregulation. Skelet Muscle. 2014 Dec 12;4(1):22. doi: 10.1186/s13395-014-0022-6. eCollection 2014. PMID 25530838
- [Background] De Palma C, Falcone S, Pisoni S, Cipolat S, Panzeri C, Pambianco S, Pisconti A, Allevi R, Bassi MT, Cossu G, Pozzan T, Moncada S, Scorrano L, Brunelli S, Clementi E. Nitric oxide inhibition of Drp1-mediated mitochondrial fission is critical for myogenic differentiation. Cell Death Differ. 2010 Nov;17(11):1684-96. doi: 10.1038/cdd.2010.48. Epub 2010 May 14. PMID 20467441
- [Background] Cordani N, Pisa V, Pozzi L, Sciorati C, Clementi E. Nitric oxide controls fat deposition in dystrophic skeletal muscle by regulating fibro-adipogenic precursor differentiation. Stem Cells. 2014 Apr;32(4):874-85. doi: 10.1002/stem.1587. PMID 24170326
- [Background] Sciorati C, Buono R, Azzoni E, Casati S, Ciuffreda P, D'Angelo G, Cattaneo D, Brunelli S, Clementi E. Co-administration of ibuprofen and nitric oxide is an effective experimental therapy for muscular dystrophy, with immediate applicability to humans. Br J Pharmacol. 2010 Jul;160(6):1550-60. doi: 10.1111/j.1476-5381.2010.00809.x. PMID 20590643
- [Background] Sciorati C, Staszewsky L, Zambelli V, Russo I, Salio M, Novelli D, Di Grigoli G, Moresco RM, Clementi E, Latini R. Ibuprofen plus isosorbide dinitrate treatment in the mdx mice ameliorates dystrophic heart structure. Pharmacol Res. 2013 Jul;73:35-43. doi: 10.1016/j.phrs.2013.04.009. Epub 2013 May 1. PMID 23644256
- [Background] D'Angelo MG, Gandossini S, Martinelli Boneschi F, Sciorati C, Bonato S, Brighina E, Comi GP, Turconi AC, Magri F, Stefanoni G, Brunelli S, Bresolin N, Cattaneo D, Clementi E. Nitric oxide donor and non steroidal anti inflammatory drugs as a therapy for muscular dystrophies: evidence from a safety study with pilot efficacy measures in adult dystrophic patients. Pharmacol Res. 2012 Apr;65(4):472-9. doi: 10.1016/j.phrs.2012.01.006. Epub 2012 Jan 25. PMID 22306844
- [Background] Cossu MV, Cattaneo D, Fucile S, Pellegrino P, Baldelli S, Cozzi V, Capetti A, Clementi E. Combined isosorbide dinitrate and ibuprofen as a novel therapy for muscular dystrophies: evidence from Phase I studies in healthy volunteers. Drug Des Devel Ther. 2014 May 2;8:411-9. doi: 10.2147/DDDT.S58803. eCollection 2014. PMID 24851040
- [Background] Sciorati C, Miglietta D, Buono R, Pisa V, Cattaneo D, Azzoni E, Brunelli S, Clementi E. A dual acting compound releasing nitric oxide (NO) and ibuprofen, NCX 320, shows significant therapeutic effects in a mouse model of muscular dystrophy. Pharmacol Res. 2011 Sep;64(3):210-7. doi: 10.1016/j.phrs.2011.05.003. Epub 2011 May 12. PMID 21609764
- [Background] Campana L, Santarella F, Esposito A, Maugeri N, Rigamonti E, Monno A, Canu T, Del Maschio A, Bianchi ME, Manfredi AA, Rovere-Querini P. Leukocyte HMGB1 is required for vessel remodeling in regenerating muscles. J Immunol. 2014 Jun 1;192(11):5257-64. doi: 10.4049/jimmunol.1300938. Epub 2014 Apr 21. PMID 24752445
- [Background] Castiglioni A, Corna G, Rigamonti E, Basso V, Vezzoli M, Monno A, Almada AE, Mondino A, Wagers AJ, Manfredi AA, Rovere-Querini P. FOXP3+ T Cells Recruited to Sites of Sterile Skeletal Muscle Injury Regulate the Fate of Satellite Cells and Guide Effective Tissue Regeneration. PLoS One. 2015 Jun 3;10(6):e0128094. doi: 10.1371/journal.pone.0128094. eCollection 2015. PMID 26039259
- [Background] Lukaski HC. Evolution of bioimpedance: a circuitous journey from estimation of physiological function to assessment of body composition and a return to clinical research. Eur J Clin Nutr. 2013 Jan;67 Suppl 1:S2-9. doi: 10.1038/ejcn.2012.149. PMID 23299867
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Yesavage, J.A., Sheikh, J.I.: 9/Geriatric Depression Scale (GDS). Clinical Gerontologist. 5, 165-173 (1986).
- [Background] Burke WJ, Roccaforte WH, Wengel SP. The short form of the Geriatric Depression Scale: a comparison with the 30-item form. J Geriatr Psychiatry Neurol. 1991 Jul-Sep;4(3):173-8. doi: 10.1177/089198879100400310. PMID 1953971
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ware J, Kosinski M, Keller SD. SF-36 physical and mental health summary scales: a user's manual. Boston, MA: The Health Institute, New England Medical Centre (1994).
- [Background] Ware JE. SF-36 Health Survey. Manual and interpretation guide. The Health Institute, New England Medical Centre. Boston, MA. 2nd ed., Nimrod Press (1997)
- [Background] Haywood KL, Garratt AM, Schmidt LJ, Mackintosh AE, Fitzpatrick R. Health Status and Quality of Life in Older People: a Structured Review of Patient-reported Health Instruments Report from the Patient- reported Health Instruments Group (formerly the Patient-assessed Health Outcomes Programme) to the Department of Health (2004).
- [Background] Irvine D, O'Brien-Pallas LL, Murray M, Cockerill R, Sidani S, Laurie-Shaw B, Lochhaas-Gerlach J. The reliability and validity of two health status measures for evaluating outcomes of home care nursing. Res Nurs Health. 2000 Feb;23(1):43-54. doi: 10.1002/(sici)1098-240x(200002)23:13.0.co;2-k. PMID 10686572
- [Background] Osborne RH, Hawthorne G, Lew EA, Gray LC. Quality of life assessment in the community-dwelling elderly: validation of the Assessment of Quality of Life (AQoL) Instrument and comparison with the SF-36. J Clin Epidemiol. 2003 Feb;56(2):138-47. doi: 10.1016/s0895-4356(02)00601-7. PMID 12654408
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Vahlberg B, Zetterberg L, Lindmark B, Hellstrom K, Cederholm T. Functional performance, nutritional status, and body composition in ambulant community-dwelling individuals 1-3 years after suffering from a cerebral infarction or intracerebral bleeding. BMC Geriatr. 2016 Feb 19;16:48. doi: 10.1186/s12877-016-0226-1. PMID 26895855